CLINICAL TRIAL: NCT00487695
Title: Confocal Laser Endomicroscopy for Improved Diagnosis of Barrett's Esophagus and Associated Neoplasia
Brief Title: Confocal Endomicroscopy for Barrett's Esophagus
Acronym: CEBE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other); Pentax, USA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: NA0002805
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Barrett's Esophagus; Esophageal Adenocarcinoma
Keywords: Barrett's esophagus; Esophageal adenocarcinoma; Endoscopy; Confocal laser endomicroscopy
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CLE followed by standard EGD (Active Comparator): Participants are randomized to have either confocal laser endomicroscopy (CLE) or standard endoscopy (EGD) first. Then 6 weeks later, they have the other procedure. This arm is for patients randomized to CLE followed by standard EGD
  Interventions: Device: confocal laser endomicroscopy (CLE); Device: standard endoscopy (EGD)
- standard EGD followed by CLE (Active Comparator): Patients are randomized to either have standard endoscopy (EGD)or confocal laser endomicroscopy (CLE) first. The second procedure is then completed 6 weeks later. This arm is for patients who had standard endoscopy first.
  Interventions: Device: confocal laser endomicroscopy (CLE); Device: standard endoscopy (EGD)

INTERVENTIONS:
Device: confocal laser endomicroscopy (CLE) — Confocal laser endomicroscopy is done by performing standard endoscopy, then using a microscope on the tip of the endoscope to obtain microscopic images of the mucosa. This is done by gently placing the tip of the endoscope on the lining of the esophagus.
  Other Names: Pentax Confocal Laser Endomicroscope(EC3870KCILK)
Device: standard endoscopy (EGD) — Standard upper endoscopy (EGD) is performed using a regular upper endoscope, which is used to look at the lining of the esophagus.
  Other Names: Olympus upper endoscope (GIF160)

SUMMARY:
The purpose of this study is to determine if confocal laser endomicroscopy (CLE) can improve detection of Barrett's esophagus, dysplasia, and early esophageal cancer.

DETAILED DESCRIPTION:
Barrett's esophagus is a leading cause of esophageal adenocarcinoma. Detection of dysplasia and early cancers in Barrett's esophagus can be challenging, time-consuming and expensive. Small lesions may be difficult to detect with standard endoscopy protocols. Confocal laser endomicroscopy (CLE) is a new type of endoscopy where a small confocal microscope is built into the tip of a standard endoscope. For this study, we are comparing confocal laser endomicroscopy (CLE) with targeted biopsies with standard endoscopy (EGD)and biopsy for Barrett's esophagus to determine if CLE is more effective for detecting dysplasia and cancer.

Participants with Barrett's esophagus in this study undergo 1) CLE with targeted mucosal biopsies (biopsy only taken if CLE shows abnormal tissue) and 2) standard EGD with biopsies. The order of procedures is randomized (some patients have CLE first while others have standard EGD first).

ELIGIBILITY:
Inclusion Criteria:

* Barrett's esophagus or suspected Barrett's-associated neoplasia
* Age > 18
* Able to give informed consent

Exclusion Criteria:

* Known advanced malignant disease
* Allergy to the fluorescent contrast agent fluorescein sodium
* Coagulopathy or bleeding disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia I Canto, MD, MHS, Principal Investigator — Division of Gastroenterology, Johns Hopkins University School of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Result] Dunbar KB, Okolo P 3rd, Montgomery E, Canto MI. Confocal laser endomicroscopy in Barrett's esophagus and endoscopically inapparent Barrett's neoplasia: a prospective, randomized, double-blind, controlled, crossover trial. Gastrointest Endosc. 2009 Oct;70(4):645-54. doi: 10.1016/j.gie.2009.02.009. Epub 2009 Jun 25. PMID 19559419

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from April 2007 to May 2008 from the gastroenterology clinics at Johns Hopkins University.
Pre-assignment Details: None of the patients enrolled were excluded prior to group assignment. 1 patient dropped out prior to the first procedure.
Groups:
- CLE Followed by Standard EGD: Patients randomized to either CLE or standard endoscopy first. The other procedure was then performed 6 weeks later. This group was randomized to CLE first, followed by standard endoscopy
- Standard EGD Followed by CLE: Patients in this group were randomized to have standard EGD followed by CLE 6 weeks later
Period: First Procedure
Arm/Group | CLE Followed by Standard EGD | Standard EGD Followed by CLE
Started | 23 | 23
Completed | 20 | 23
Not Completed | 3 | 0
Not completed — invasive cancer on EGD (excl criteria) | 1 | 0
Not completed — active wheezing (did not have procedure) | 1 | 0
Not completed — esophageal stricture found (excl crit) | 1 | 0
Period: Second Procedure
Arm/Group | CLE Followed by Standard EGD | Standard EGD Followed by CLE
Started | 20 | 23
Completed | 19 | 20
Not Completed | 1 | 3
Not completed — active wheezing | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Patients received both procedures (CLE and standard EGD), so baseline characteristics are reported for the group
Arm/Group | All Study Participants
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Yield for Neoplasia in High Risk Patients(Suspected Neoplasia)
Description: The yield for neoplasia is calculated by the number of biopsies showing neoplasia over the total number of biopsies taken (normal + neoplastic biopsies)
Time Frame: 6 weeks
Population: Analysis was per protocol as the patients who did not undergo CLE could not be analyzed at all (cannot compare 2 procedures when only one (or zero) are performed. This analysis looks specifically at patients with Barrett's and suspected (but not known) neoplasia.
Measure: Number; unit: percent yield for neoplasia
Groups:
- Confocal Laser Endomicroscopy; Standard Endoscopy: all patients had both confocal endomicroscopy and standard endoscopy in crossover fashion. For outcome, will compare the results of CLE and standard endoscopy.
Arm/Group | Confocal Laser Endomicroscopy | Standard Endoscopy
Number analyzed (Participants) | 16 | 16
percent yield for neoplasia | 34 (0) | 17 (0)
Statistical Analysis 1: Comparison: Confocal Laser Endomicroscopy vs Standard Endoscopy; Our hypothesis was that the yield for neoplasia would be higher using confocal laser endomicroscopy compared to standard endoscopy. The null hypothesis would be that there is no difference in yield for neoplasia when CLE is used compared to standard endoscopy. We estimated that the yield for neoplasia would increase from 10% to 40% using CLE and the calculated sample size was 37. We planned to enroll 48 patients to allow for possible dropouts; Test type: Superiority or Other; p = 0.01, Wilcoxon signed rank

2. Secondary Outcome: Mean Number of Biopsies With Neoplasia in High Risk Patients (Suspected Neoplasia)
Description: The number of biopsies from each procedure (i.e. biopsies taken during CLE, or biopsies taken during standard EGD) that showed neoplasia. Neoplasia is high grade dysplasia or cancer. This analysis looks at patients with Barrett's suspected (but not known) neoplasia.
Time Frame: 6 weeks
Population: Analysis was per protocol. Each participant was compared to self, so if the participant did not complete the study, no comparison could be made.
Measure: Mean (Full Range); unit: mean number of biopsies with neoplasia
Arm/Group | Confocal Laser Endomicroscopy | Standard Endoscopy
Number analyzed (Participants) | 16 | 16
mean number of biopsies with neoplasia | 3.1 [0 to 15] | 3.7 [0 to 19]
Statistical Analysis 1: Comparison: Confocal Laser Endomicroscopy vs Standard Endoscopy; The number of biopsies showing neoplasia was determined for each procedure (confocal laser endomicroscopy, standard EGD). These were compared; Test type: Superiority or Other; p = 0.89, Wilcoxon signed-rank

3. Secondary Outcome: Mean Number of Biopsies Taken in High Risk Patients (Suspected Neoplasia)
Description: The number of biopsies taken during each procedure (i.e. the number of biopsies taken during CLE, or the number of biopsies taken during standard EGD). Biopsies are taken during CLE only if CLE shows that the esophageal mucosa is abnormal. Esophageal biopsies are taken during standard EGD using a standard Barrett's esophagus protocol (4 quadrants, every 1-2 cm of the Barrett's esophagus). This analysis looks at the Barrett's patients with suspected (but not known) neoplasia.
Time Frame: 6 weeks
Population: per protocol as participants would only have data to compare if they completed both endoscopies
Measure: Mean (Full Range); unit: mean number of biopsies
Arm/Group | Confocal Laser Endomicroscopy | Standard Endoscopy
Number analyzed (Participants) | 16 | 16
mean number of biopsies | 9.8 [1 to 22] | 23.7 [3 to 41]
Statistical Analysis 1: Comparison: Confocal Laser Endomicroscopy vs Standard Endoscopy; The null hypothesis would be that CLE does not decrease the number of biopsies needed to make a diagnosis compared to standard endoscopy; Test type: Superiority or Other; p = 0.002, wilcoxon signed rank test

4. Secondary Outcome: Diagnostic Yield for Neoplasia in Barrett's Surveillance Patients
Description: Our hypothesis was that the yield for neoplasia would be higher using confocal laser endomicroscopy compared to standard endoscopy. The null hypothesis would be that there is no difference in yield for neoplasia when CLE is used compared to standard endoscopy. This analysis looks specifically at patients who were referred for surveillance of Barrett's esophagus (no suspected neoplasia).
Time Frame: 6 weeks
Population: Analysis was per protocol as the patients who did not undergo CLE could not be analyzed at all (cannot compare 2 procedures when only one (or zero) are performed).
Measure: Number; unit: percent yield for neoplasia
Arm/Group | Confocal Laser Endomicroscopy | Standard Endoscopy
Number analyzed (Participants) | 23 | 23
percent yield for neoplasia | 0 | 0

5. Secondary Outcome: Mean Number of Biopsies With Neoplasia in Barrett's Surveillance Patients
Description: The number of biopsies from each procedure (i.e. biopsies taken during CLE, or biopsies taken during standard EGD) that showed neoplasia. Neoplasia is high grade dysplasia or cancer. This analysis looks at patients undergoing surveillance EGD for Barrett's esophagus (no suspected neoplasia).
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Mean (Full Range); unit: number of biopsies with neoplasia
Arm/Group | Confocal Laser Endomicroscopy | Standard Endoscopy
Number analyzed (Participants) | 23 | 23
number of biopsies with neoplasia | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Confocal Laser Endomicroscopy vs Standard Endoscopy; The number of biopsies showing neoplasia was determined for each procedure (confocal laser endomicroscopy, standard EGD). These were compared. This analysis looks at the patients referred for Barrett's surveillance EGD (no suspected neoplasia); Test type: Superiority or Other; p = 1.0, Wilcoxon signed-rank

6. Secondary Outcome: Mean Number of Biopsies Taken in Barrett's Surveillance Patients
Description: The number of biopsies taken during each procedure (i.e. the number of biopsies taken during CLE, or the number of biopsies taken during standard EGD). Biopsies are taken during CLE only if CLE shows that the esophageal mucosa is abnormal. Esophageal biopsies are taken during standard EGD using a standard Barrett's esophagus protocol (4 quadrants, every 1-2 cm of the Barrett's esophagus). This analysis looks at the patients with Barrett's esophagus in the study who were undergoing surveillance EGD (no suspected neoplasia).
Time Frame: 6 weeks
Population: Analysis was per protocol. Each participant was compared to self, so if the participant did not complete, the study, no comparison could be made. The patients in this analysis were referred for surveillance of Barrett's esophagus (no suspected neoplasia).
Measure: Mean (Full Range); unit: mean number of biopsies
Arm/Group | Confocal Laser Endomicroscopy | Standard Endoscopy
Number analyzed (Participants) | 23 | 23
mean number of biopsies | 1.7 [0 to 12] | 12.6 [1 to 28]
Statistical Analysis 1: Comparison: Confocal Laser Endomicroscopy vs Standard Endoscopy; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank

ADVERSE EVENTS:
Time Frame: Adverse event data was collected after each procedure and for an average of one month after the last procedure.
Groups:
- Confocal Laser Endomicroscopy; Standard EGD: Adverse even reporting is being done by procedure type (ie confocal laser endomicroscopy vs. standard endoscopy)
Arm/Group | Confocal Laser Endomicroscopy | Standard EGD
Serious Adverse Events (participants affected / at risk) | 1/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Confocal Laser Endomicroscopy (N=39) | Standard EGD (N=39)
post-procedure pneumonia (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Relatively small study (39 patients) and performed at a tertiary care, referral center, which can reduce generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No